CLINICAL TRIAL: NCT06181136
Title: A Phase 1/2, Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DNL126 in Pediatric Participants With Mucopolysaccharidosis Type IIIA (Sanfilippo Syndrome Type A)
Brief Title: Study of DNL126 in Pediatric Participants With Mucopolysaccharidosis Type IIIA (Sanfilippo Syndrome Type A)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DNLI-I-0001
Record Dates: First submitted 2023-12-04; First posted 2023-12-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Mucopolysaccharidosis Type IIIA
Keywords: Sanfilippo Syndrome; MPS IIIA
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A1 (Experimental): Participants with MPS IIIA
  Interventions: Drug: DNL126
- Cohort A2 (Experimental): Participants with MPS IIIA
  Interventions: Drug: DNL126
- Cohort A3 (Experimental): Participants with MPS IIIA
  Interventions: Drug: DNL126
- Cohort B1 (Experimental): Participants with MPS IIIA
  Interventions: Drug: DNL126
- Cohort B2 (Experimental): Participants with MPS IIIA
  Interventions: Drug: DNL126

INTERVENTIONS:
Drug: DNL126 — intravenous repeating dose

SUMMARY:
This is a multicenter, open-label, Phase 1/2 study to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and clinical efficacy of DNL126 in participants with Sanfilippo syndrome Type A (MPS IIIA). The core study period is 25 weeks (approximately 6 months); followed by an open-label extension (OLE), which extends through Week 97 (approximately 18 months); and a long-term extension (LTE), which extends through Week 193 (Year 4). Participants with MPS IIIA will be enrolled in two planned cohorts, and additional participants with MPS IIIA may be enrolled in three optional cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of MPS IIIA
* For Cohort A2: No more than 1 participant may have predictors of a slow-progressing phenotype
* For Cohort A3: Approximately 2 participants will have predictors of the slow-progressing phenotype
* For Cohort B1: Have a severe phenotype based on having at least one of the following:

  * An older sibling with the same genotype and severe MPS IIIA, in the opinion of the investigator
  * A definitive genotype indicative of severe MPS IIIA, in the opinion of the investigator
  * Clinical symptoms of MPS IIIA prior to 28 months of age that, in the opinion of the investigator, are indicative of severe MPS IIIA
* For Cohort B2: Are an older sibling of a participant in Cohort B1 (who has already been confirmed to be eligible for dosing) with MPS IIIA, the same causative genotype, and who has severe MPS IIIA in the opinion of the investigator

Key Exclusion Criteria:

* Have unstable or poorly controlled medical condition(s) or significant medical or psychological comorbidity or comorbidities that, in the opinion of the investigator, would interfere with safe participation in the trial or interpretation of study assessments
* Have lost the ability to walk independently, in the opinion of the investigator
* Are unable to take the majority of nutrition via mouth, in the opinion of the investigator
* For Cohort B only: Are homozygous or compound heterozygous for the N-sulfoglucosamine sulfohydrolase (SGSH) S298P mutation or any other mutation known to be associated with slow-progressing phenotype
* Have used any CNS-targeted MPS IIIA enzyme replacement therapy (ERT) (eg, intrathecal SGSH or TfR-mediated SGSH delivery to CNS) within 3 months before Day 1
* Have a prior history of hematopoietic stem cell transplantation
* Have a prior history of gene therapy
* Have used genistein or anakinra within 7 days of screening or intended use of genistein or anakinra during the study
* Have a documented likely pathogenic mutation sufficient to cause disease (eg, taking into account zygosity) of other genes that are known to be associated with developmental delay, seizures, or other significant CNS disorders
* Have clinically significant thrombocytopenia, other clinically significant coagulation abnormality, significant active bleeding, or require treatment with an anticoagulant or more than two antiplatelet agents
* Contraindication for lumbar punctures
* Contraindication for MRI scan
* Have a clinically significant history of stroke, status epilepticus, head trauma with loss of consciousness, or any clinically significant CNS disease that is not MPS IIIA-related within 3 months of screening
* Have had a ventriculoperitoneal (VP) shunt placed or a clinically significant VP shunt malfunction within 30 days of screening
* Have any clinically significant CNS trauma or disorder, including severe untreated intracranial hypertension or brain surgery, that, in the opinion of the investigator, may interfere with assessment of study endpoints or make participation in the study unsafe

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in cerebrospinal fluid (CSF) concentration of heparan sulfate (HS) | 49 weeks

SECONDARY OUTCOMES:
Percentage change from baseline in urine concentration of HS (normalized to creatinine) | 49 weeks
Change from baseline in liver volume | 49 weeks
Percentage change from baseline in serum neurofilament light chain (NfL) concentration | 73 weeks
Participants with CSF HS concentration within the normal range | 49 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Claire Meyer, MD, Study Director — Denali Therapeutics
Locations (4):
- United States (4):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Baylor College of Medicine and Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No